CLINICAL TRIAL: NCT04004949
Title: The Effect of Scapular Dyskinesia on the Scapular Balance Angle & Upper Extremity Sensorimotor Function in Stroke Patients With Spasticity
Brief Title: the Effect of Scapular Dyskinesia on the Scapular Balance Angle & Upper Extremity Sensorimotor Function in Spastic Stroke Patient. The Patients Were Diagnosed With the Lateral Scapular Slide Test, Fugl-Meyer Upper Extremity (FMUE) Scale Scores & Scapular Balance Angle Test (SBA).
Status: Completed | Type: Observational
Sponsor: Lama Saad El-Din Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Lama Saad El-Din Mahmoud, lecturer of neurology & neurosurgery for physical therapy, October 6 University
Organization: October 6 University (Other)
Other Study IDs: 12341234
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Post Stroke Scapular Dyskinesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group (high scapular dyskinesia ): group A (30 patients): with high scapular dyskinesia scores
  Interventions: Other: Assessment of scapular balance angle and upper extremity sensorimotor function
- control group (low or no scapular dyskinesia ): group B (30 patients): with low or no scapular dyskinesia scores. (30 patients): with low or no scapular dyskinesia scores.
  Interventions: Other: Assessment of scapular balance angle and upper extremity sensorimotor function

INTERVENTIONS:
Other: Assessment of scapular balance angle and upper extremity sensorimotor function — The patients were diagnosed with the Lateral scapular slide test using Palpation meter (PALM) device, Fugl-Meyer upper extremity (FMUE) Scale scores & scapular balance angle test (SBA).

SUMMARY:
to investigate the effect of Scapular dyskinesia on the scapular balance angle & upper extremity Sensorimotor Function in spastic stroke patient.

DETAILED DESCRIPTION:
Background: Post stroke Scapular dyskinesia leads to scapulohumeral pain & dysfunction were associated with decreased motor function, somatosensory function, limited range of motion, and spasticity.

Objective: to investigate the effect of Scapular dyskinesia on the scapular balance angle & upper extremity Sensorimotor Function in spastic stroke patient.

Methods: sixty patients from both sexes were participated in this study. All the patients were diagnosed as spastic stroke patients. The patients were divided into two equal groups; group A (30 patients): with high scapular dyskinesia scores, group B (30 patients): with low or no scapular dyskinesia scores. The patients were diagnosed with the Lateral scapular slide test using Palpation meter (PALM) device, Fugl-Meyer upper extremity (FMUE) Scale scores & scapular balance angle test (SBA).

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed as stroke patient
* stroke onset at least 5 months prior to study enrollment and
* decreased sensorimotor function in the affected arm, but ability to use the arm to some extent in daily activities with functional to subfunctional manual muscle test
* age ranged from 35:50
* both sexes

Exclusion Criteria:

* difficulty to communicate or to understand test instructions
* other conditions that caused pain (for example fibromyalgia and arthritis)
* severe depression or other psychiatric symptoms
* patient with other upper limb musculoskeletal problems

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sixty stroke patients were randomly selected from Kasr El-Aini Neurological Department, outpatient clinic of Faculty of Physical Therapy, Cairo University, October 6 university hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
the Lateral scapular slide test | 1 day
  for the measurement of scapular dyskinesia, the Lateral scapular slide test using Palpation meter (PALM) device,
  marked inferior angles of scapula and the other arm was moved to reach the marked corresponding spinous process Both sides' readings were recorded and the differences between them were calculated
  Bilateral difference of 1.5 cm considered the threshold for deciding whether scapular asymmetry is abnormal A distance 1.5 cm greater than the contralateral side in any position suggests scapulothoracic weakness with secondary scapulothoracic protraction
Fugl-Meyer Assessment (FMA) scale | 1 day
  Fugl-Meyer upper extremity (FMUE) Scale scores is an index to assess the sensorimotor impairment in individuals who had stroke.
  The motor section score ranges from 0 to 66, and the score related to exteroceptive and proprioceptive sensitivity ranges from 0 to 12. The lowest and highest scores correspond to worse and better function, respectively FMUE Scale scores < 31 corresponded with 'no to poor' upper extremity capacity, while 32 to 47 represented 'limited capacity', 48 to 52 represented 'notable capacity' and 53 to 66 represented 'full' upper extremity capacity
scapular balance angle (SBA): | 1 day
  for Measurement of scapular balance angle
  The inferior angle of the scapula was marked bilaterally and a line was drawn connecting these marks. Another vertical line between C7 and T10 spinous processes was drawn. The angles formed by the line joining both inferior angles of the scapula with the vertical line running through the spine were measured (The difference between these two angles corresponded to the scapular balance angle The values for the SBA in healthy population were 2.505±2.340° while the abnormality criteria were with an angle greater than 7.185°

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, Giza, El-Sheikh Zayed City Giza 1133 Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
publication research study